CLINICAL TRIAL: NCT07223437
Title: REVASC-PAD: REstricted VASCular Exercise for Peripheral Arterial Disease - A Feasibility Study at University of Tennessee Medical Center
Acronym: REVASC-PAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5460; Institutional Review Board (Other: The University of Tennessee Health Science Center)
Record Dates: First submitted 2025-10-24; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blood Flow Restriction (BFR) Training (Experimental): Participants perform supervised lower-body resistance training using pneumatic cuffs (Smart Cuff Pro or equivalent) applied to the proximal thighs. Cuffs are inflated to 60-80% of the participant's measured arterial occlusion pressure (AOP). Pressure is increased at Weeks 5 and 9 based on tolerance. Cuff inflation will not exceed 80% of limb occlusion pressure. Cuffs will be immediately deflated if participants' vitals suggest poor tolerance.
  Interventions: Behavioral: Blood Flow Restriction Cuff System
- Low-Load Traditional Resistance Training (LL-RT) (Active Comparator): Participants perform the same two calf exercises (seated and standing calf raises) without BFR cuffs. If participants demonstrate the ability to complete all prescribed repetitions without undue strain, planned load progressions of approximately 5-10% 1RM will be introduced at Weeks 5 and 9. Repetitions and sets will remain fixed to match the BFR protocol.
  Interventions: Behavioral: Low-load Resistance Training
- High-Load Traditional Resistance Training (HL-RT) (Active Comparator): Participants in this group will perform seated and standing calf raises following a more conventional strength training model. Similar to the other groups, if participants can complete their prescribed workload without excessive strain, two planned load progressions (5-10% 1RM) will be applied at Weeks 5 and 9. Repetitions and sets will remain fixed to preserve consistency in training structure across groups. This group serves as a benchmark for conventional resistance training in clinical and musculoskeletal rehabilitation populations.
  Interventions: Behavioral: High-load Resistance Training

INTERVENTIONS:
Behavioral: Blood Flow Restriction Cuff System — All BFR resistance sessions will include two standardized lower-extremity exercises: seated calf raises and standing calf raises. Each session will follow this protocol:
  1. 1 set of 30 repetitions, followed by 3 sets of 15 repetitions
  2. 30 seconds rest between sets, with the cuff remaining inflated
  3. Load set at 20-35% of 1RM
  4. Cuff deflated immediately after the fourth set or after 6 continuous minutes of inflation, whichever comes first
  Arms: Blood Flow Restriction (BFR) Training
Behavioral: Low-load Resistance Training — Two resistance exercises (seated and standing calf raises) using the same repetition structure
  1. 1 set of 30 repetitions, followed by 3 sets of 15 repetitions
  2. Load set at 20-35% of 1RM
  3. 30 seconds rest between sets
  4. No BFR cuffs will be used
  Arms: Low-Load Traditional Resistance Training (LL-RT)
Behavioral: High-load Resistance Training — Each session includes:
  1. 3 sets of 8-12 repetitions
  2. Load set at 60-70% of 1RM
  3. Rest periods of 60-90 seconds between sets
  4. No BFR cuffs will be used
  Arms: High-Load Traditional Resistance Training (HL-RT)

SUMMARY:
The purpose of this study is to evaluate the effects of Blood Flow Restriction (BFR) training on walking function, health-related quality of life, and safety among adults with Peripheral Arterial Disease (PAD).

The main aims of the study are:

1. Evaluate change in walking function among patients with PAD undergoing BFR training. The investigators will assess change in Six-Minute Walk Test (6MWT) distance from baseline to post-intervention and 3-month follow-up to compare functional improvements between the BFR group and the two control groups
2. Assess changes in health-related quality of life among patients with PAD undergoing BFR training. The investigators will use the EuroQol 5-Dimension 5-Level (EQ-5D-5L) scale to evaluate quality-of-life changes from baseline to post-intervention and 3-month follow-up across all study arms
3. Evaluate the safety and feasibility of a supervised BFR training program for patients with PAD. The investigators will compare adverse event (AE) and serious adverse event (SAE) rates across study arms, while also monitoring sessional ratings of perceived exertion (RPE), dyspnea, and claudication pain as indicators of symptom response and exercise tolerance. Feasibility will be assessed through enrollment success, intervention adherence, and retention rates across groups

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Diagnosed peripheral arterial disease with stable claudication (symptomatic presentation unchanged for 6 months)
3. Ankle-brachial index (ABI) between 0.4 and 0.9.
4. Eligible referral to cardiovascular or pulmonary rehabilitation
5. Prior revascularization permitted if symptoms are stable and other criteria are met

Exclusion Criteria:

1. Recent change in resting ECG suggesting significant ischemia, recent myocardial infarction (within 2 weeks), or another acute cardiac event
2. Unstable angina
3. Uncontrolled cardiac arrhythmias
4. Symptomatic severe aortic stenosis or other significant valvular disease
5. Decompensated symptomatic heart failure
6. Acute pulmonary embolism or infarction
7. Acute noncardiac disorder likely to interfere with or be worsened by exercise (e.g., infection, thyrotoxicosis)
8. Acute myocarditis or pericarditis
9. Acute thrombophlebitis
10. Physical disability precluding safe or adequate exercise performance
11. Significant electrolyte abnormalities
12. Clinically significant tachyarrhythmias or bradyarrhythmias
13. High-degree atrioventricular block
14. Atrial fibrillation with uncontrolled ventricular response
15. Hypertrophic obstructive cardiomyopathy with resting left ventricular outflow gradient of >25 mmHg
16. Known active aortic dissection
17. Severe resting arterial hypertension (SBP>200mmHg or DBP >110 mmHg)
18. Mental impairment preventing cooperation with study procedures
19. Current pregnancy
20. Moderate to severe peripheral neuropathy
21. Open wounds or compromised skin near BFR cuff site
22. Active DVT or thromboembolic event within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-11-05 (Estimated); Primary Completion 2027-11-05 (Estimated); Study Completion 2027-11-05 (Estimated)

PRIMARY OUTCOMES:
Walking Function | Baseline (Visit 1), post-intervention (8 to 12 weeks), and 3-month follow-up (3MF)
  Change in walking distance measured by the Six-Minute Walk Test (6MWT) from baseline to end of intervention and 3-month follow-up visit.
Quality of Life (QoL) (1) | Baseline (Visit 1), post-intervention (8 to 12 weeks), and 3-month follow-up (3MF)
  Change in health-related quality of life as assessed by EuroQol 5-Dimension 5-Level (EQ-5D-5L) from baseline to post-intervention and 3-month follow-up
Quality of Life (QoL) (2) | Baseline (Visit 1), post-intervention (8 to 12 weeks), and 3-month follow-up (3MF)
  Change in depressive symptoms as assessed by Patient Health Questionnaire-9 (PHQ-9) from baseline to post-intervention and 3-month follow-up
Quality of Life (QoL) (3) | Baseline (Visit 1), post-intervention (8 to 12 weeks), and 3-month follow-up (3MF)
  Change in self-reported walking function and symptom burden assessed by using REVASC-PAD Walking Questionnaire from baseline to post-intervention and 3-month follow-up

SECONDARY OUTCOMES:
Claudication Onset Time (COT) during 6MWT | Baseline, post-intervention (8 to 12 weeks), and 3 months post-intervention
  Time to onset of claudication symptoms during 6MWT at baseline, post-intervention, and 3-month follow-up
Ratings of Perceived Exertion (RPE), Dyspnea, and Claudication Pain | Multiple assessments from Visit 2 through end of intervention (approximately 8 to 12 weeks)
  Session-based self-reported symptom ratings collected at each supervised exercise session from Visit 2 to end of intervention (approximately 8 to 12 weeks). These ratings assess exercise tolerance and symptom burden during blood flow restriction training.
Adverse Event (AE) and Serious Adverse Event (SAE) Rates | Baseline to 3-month follow-up
  Number and rate of adverse events and serious adverse events occurring during the study period.
Enrollment, Retention, and Adherence Rates | Baseline to 3-month follow-up
  Rates of successful enrollment, participant retention at post-intervention and 3-month follow-up, and adherence to prescribed exercise sessions

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States